# PHASE 2 EFFICACY & SAFETY EVALUATION OF ADVANTAGE ANTI-CARIES VARNISH FOR PRIMARY PREVENTION

Study Acronym: NGIHN SERI MWAHU

**Advantage Protocol Number: 2019-10-19** 

**Clinical Trial Registration Number: NCT04947527** 

IND #128835

IND Sponsor: Advantage Silver Dental Arrest, LLC PO Box 12746 Salem, OR 97309-0746

**Sponsor Contact:** Peter Milgrom, DDS

Principal Investigator: Ohnmar Tut, BDS MPhil

Medical Monitor: John Hedson, MD

**Regulatory Monitors:** Douglas Bierer, PhD

**Version Number: 2.4** 

**Version Date:** 07/01/2022

| Protocol # 2019-10-19 | Version 2.4 / July 1, 202 |
|---|---|
| F10t0c0t# 2019-10-19 | Version 2.47 July 1, 202 |
| PROTOCOL APPROVAL | |
| Phase 2 Efficacy & Safety Evaluation of Advanta | age Anti-Caries Varnish for Primary Prevention |
| STUDY ACRONYM: | NGIHN SERI MWAHU |
| Ohnmar K. Tut, BDS MPhil | Date |
| Principal Investigator | Date |
| Peter Milgrom, DDS | Date |
| Sub-Investigator | Date |

Version 2.4 / July 1, 2022

# STATEMENT OF COMPLIANCE

The study will be carried out in accordance with Good Clinical Practice (GCP) as required by the following:

- United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, and 21 CFR Part 312)
- ICH E6; 62 Federal Register 25691 (May 9, 1997)

All key personnel (all individuals responsible for the design and conduct of this study) have completed Human Subjects Protection Training.

#### Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention

Protocol # 2019-10-19


#### **SIGNATURE PAGE**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable US federal regulations and ICH guidelines.

I have carefully read this protocol, and agree that it contains all the necessary information for conducting the study safely.

I will conduct this study in strict accordance with this protocol and according to the current Good Clinical Practice (GCP) regulations and guidelines [21 CFR (Code of Federal Regulations) Parts 11, 50, 54 and 56 and ICH (International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use) Topic E6 (R1)], and local regulatory requirements. Any changes in procedure will only be made if necessary to eliminate immediate hazards and/or to protect the safety, rights or welfare of subjects.

I will provide copies of the protocol and all other information relating to the pre-clinical and prior clinical experience, which were furnished to me, to all physicians and other study personnel responsible to me who participate in this study. I will discuss this information with them to assure that they are adequately informed regarding the study drug and conduct of the study.

I will ensure that the drugs supplied to me for this study will be used only for administration to subjects enrolled in this study protocol and for no other purpose.

I agree to keep records on all subject information (case report forms, informed consent statements, drug accountability records, and all other information collected during the study) in accordance with the current GCP, local and national regulations.

| Date | |
|------|------|
| _ | Date |

| Protocol # 2019-10-19 | Version 2.4 / July 1, 202 |
|-----------------------|---------------------------|
| SUMMARY OF CHANGES | |
| Protocol Amendments | |

# **TABLE OF CONTENTS**

| PROTOCOL APPROVAL | 2 |
|---|---|
| STATEMENT OF COMPLIANCE | 3 |
| SIGNATURE PAGE | 4 |
| SUMMARY OF CHANGES | 5 |
| Protocol Amendments | 5 |
| LIST OF ABBREVIATIONS | 10 |
| PROTOCOL SUMMARY | 11 |
| Alignment with ICH Topic E 5 (R1) [Ethnic Factors in the Acceptability o Clinical Data] | |
| SCHEMATIC OF STUDY DESIGN | 14 |
| 1. Key Roles | 15 |
| 2. Introduction: Background Information and Scientific Rationale | 16 |
| 2.1 Background Information | 16 |
| 2.2.1 Potential Risks and Benefits 2.2.1 Potential Risks 2.2.2 Known Potential Benefits | 18 |
| 3. Objectives | 19 |
| 3.1 Study Objectives | 19 |
| 3.2.1 Primary Outcome Measures | 19 |
| 4. Study Design | 19 |
| 4.1 Rationale for Study Design | 19 |
| 4.2 Rationale for Dosage | 20 |
| 5. Study Enrollment and Withdrawal | 20 |
| 5.1 Subject Numbers | 20 |
| 5.2 Subject Inclusion Criteria | |
| 5.3 Subject Exclusion Criteria | |
| 5.4 Discussion of Subject Characteristics | |
| 5.5 Strategies for Recruitment and Retention | 21 |

| | | Treatment Assignment Procedures | |
|---|---|---|---|
| | • | 6.1 Subject Identification Numbers | |
| | <b>5.7</b> | Masking Procedures | |
| | | • | |
| | <b>5.8</b><br>5.8 | Reasons for Withdrawal | |
| | 5.9 | Termination of Study | 23 |
| 6. | Invest | tigational Product | 24 |
| | 6.1 | Investigational Product Description | 24 |
| | 6. | 1.1 Acquisition | 24 |
| | _ | 1.2 Formulation, Packaging, and Labeling | |
| | 6.2 | Dosage, Preparation and Administration of Study Investigational Products | 25 |
| | 6.3 | Accountability Procedures for the Investigational Product(s) | 25 |
| | 6.4 | Assessment of Subject Compliance with Investigational Product | 25 |
| | 6.5 | Coding/Emergency Treatment Disclosure | 25 |
| | 6.6 | Concomitant Medications/Treatments | 26 |
| 7. | Study | Schedule/Procedures and Evaluations | 26 |
| | 7.1 | Subject recruitment procedures: | 26 |
| | 7.2 | Baseline Visit | 27 |
| | 7.3 | Visits 2-8 Treatment Visit | 27 |
| | 7.4 | Visit 9 Year 2 Exam Visit | 28 |
| | 7.5 | Premature Withdrawal | 28 |
| | 7.6 | Unscheduled Visit | 28 |
| 8. | Asses | ssments | 29 |
| | 8.1 | Primary and Secondary Outcome Variables | 29 |
| | | Efficacy Assessments | |
| | | 2.1 Caries Examination | |
| | | Safety Assessments | |
| 9. | Asses | ssment of Safety | 30 |
| | 9.1 | Specification of Safety Parameters | 30 |
| | 9.2 | Methods and Timing for Assessing, Recording, and Analyzing Safety | |
| | ⊦arame | ters | 30 |

| | 9.3 Adverse Events | 30 |
|---|---|---|
| | 9.4 Expected Adverse Reactions | 31 |
| | 9.5 Serious Adverse Events | 31 |
| | 9.5.1 Unanticipated Problems | |
| | 9.5.2 Procedures to be Followed in the Event of Abnormal Clinical Findings | 32 |
| | 9.6 Reporting Procedures | 32 |
| | 9.6.1 Reportable Events | |
| | 9.6.2 Serious Adverse Events | |
| | 9.6.3 Adverse Event Causality Definitions | |
| | 9.6.4 Adverse Event Severity Definitions | 34 |
| | 9.7 Responsibilities of Investigator/Sponsor for Reporting SAEs | |
| | 9.7.1 Regulatory Reporting for Studies Conducted Under an IND | |
| | 9.7.2 Other Unanticipated Problems | 34 |
| | 9.8 Type and Duration of Follow-up of Subjects after Adverse Events | 35 |
| | 9.9 Halting Rules | 35 |
| 10. | Site Monitoring | |
| | 10.1 Clinical Site Monitoring | |
| | • | |
| | 10.2 Regulatory Inspections | |
| 11. | Statistical Considerations | 36 |
| | 11.1 Study Hypotheses | 36 |
| | 11.2 Sample Size Considerations | 36 |
| | 11.3 Statistical Analysis Plan | 37 |
| | 11.3.1 Primary Statistical Analysis. | |
| | 11.3.2 Analysis of Safety Data. | |
| | 11.3.3 Participant Disposition. | 38 |
| 12. | Source Documents and Access to Source Data/Documents | <i>38</i> |
| | 12.1 Primary Source Documents | 38 |
| | 12.2 CRF Worksheets | 38 |
| 13. | Ethics/Protection of Human Subjects | 39 |
| | 13.1 Ethical Standard | 39 |
| | 13.2 Institutional Review Board | 39 |
| | 13.3 Amendments | 39 |
| | 13.4 Informed Consent Process | 39 |
| | 13.5 Exclusion of Women, Minorities, and Children (Special Populations) | 40 |

# Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention

| | 1+ | റററി | -44 | 20 | 40 | 1 | ^ | 11 | _ |
|---|------|------|-----|-----|----|----|------|----|---|
| Н | 'not | ററവ | # | 7() | 19 | -1 | ( )- | 13 | ٧ |


| | 13.6 Subject Confidentiality | 40 |
|-----|---------------------------------------|----------|
| | 13.7 Study Discontinuation | 40 |
| 14. | Data Handling and Record Keeping | 40 |
| | 14.1 Data Management Responsibilities | 40 |
| | 14.2 Data Capture Methods | 41 |
| | 14.3 Types of Data | 41 |
| | 14.4 Timing/Reports | 41 |
| | 14.5 Study Records | |
| | 14.5.1 Study File and Site Documents | 42<br>43 |
| | 14.6 Protocol Deviations | |
| 14. | 7 Protocol Violations | |
| | Publication Policy | |
| | Literature References | |
| 17. | Addendum | 47 |


# LIST OF ABBREVIATIONS

AE Adverse Event/Adverse Experience

ADA American Dental Association CFR Code of Federal Regulations

CRF Case Report Form

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

ICF Informed Consent Form

ICH International Conference on Harmonization

ICMJE International Committee of Medical Journal Editors

IND Investigational New Drug Application

IRB Institutional Review Board

MedDRA<sup>®</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures NDA New Drug Application

OHRP Office for Human Research Protections

PCP Primary Care Physician
PHI Protected Health Information

PI Principal Investigator

10% PVPI 10% Povidone/1.0% Iodine SAE Serious Adverse Event

S-ECC Severe Early Childhood Caries
SOP Standard Operating Procedure
WIRB Western Institutional Review Board

WCG IRB WIRB-Copernicus Group Institutional Review Board

# **PROTOCOL SUMMARY**

| Title | Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention Acronym Title: NGIHN SERI MWAHU |
|---|---|
| Précis | The purpose of the study is to determine the efficacy & safety of |
| | Advantage Anti-Caries Varnish for primary prevention |
| Objectives | Primary To determine if Advantage Anti-Caries Varnish (test varnish) is superior to an active control varnish (5% NaF, no PVP-I) in the prevention of caries lesions in the primary dentition. Specifically, prevention of caries lesions in primary teeth that either are sound, have only d <sub>1</sub> (white spots) lesions or unerupted at baseline. Secondary To document the safety of the test varnish. |
| | , |
| Study Population | Children 6 to 24 months at time of entry, approximately 50% male, 50% female |
| Phase | 2 |
| Number of Sites | One: Pohnpei State, Federated States of Micronesia |
| Study Duration | The entire study duration will be about 3 years, allowing for start-up, training, the active phase, and close out. |
| Subject<br>Participation<br>Duration | The total duration of subject participation is 24 months. |
| Description of Agent or Intervention | Single-center, double-blind, controlled Phase 2 study with parallel groups of children. Subjects will be randomized to receive either test varnish or control varnish topically to the teeth. Treatment will be administered quarterly for up to 24 months. |
| Estimated Time to<br>Complete<br>Enrollment | 3 months |
| Number of Subjects | Total number of subjects planned is: 254 |
| Inclusion Criteria | <ol> <li>The subject's parent or legal guardian must provide signed dated informed consent (parent permission form).</li> <li>The subject's parent or legal guardian must be willing and abl comply with study requirements.</li> <li>The subject is aged 6 to 24 months at the time of the enrollment.</li> <li>The subject must be in good general health as evidenced by pareport.</li> </ol> |

# Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention

Protocol # 2019-10-19


| | 5. The subject will have at least 1 erupted tooth that is either sound or has only a d <sub>1</sub> (white spots) lesion. |
|---|---|
| Exclusion Criteria | <ol> <li>Previous treatment with fluoride varnish</li> <li>Known allergy to iodine</li> <li>Diagnosis of thyroid disease</li> <li>Chronic, prophylactic use of antibiotics</li> <li>Treatment with another investigational drug or other intervention within 30 days preceding the Baseline Visit.</li> <li>Visible cavities (d<sub>2-4</sub>) in the erupted primary teeth</li> <li>Presence of intraoral soft tissue pathology</li> <li>Parent anticipates the child will move from Pohnpei during the next 2 years.</li> </ol> |
| Route and Dosage<br>Form | Treatment applied to teeth topically (0.2 mL test or control) |
| Primary Outcome<br>Measures | Efficacy: Primary: New surface-level primary caries (d <sub>2-4</sub> mfs) at 24-months post baseline Secondary: Presence/Absence of new caries (d <sub>2-4</sub> mfs) at 12-months post baseline |
| Secondary<br>Outcome Measures | Safety: Adverse event occurrence |


# Alignment with ICH Topic E 5 (R1) [Ethnic Factors in the Acceptability of Foreign Clinical Data]

Alignment with ICH Topic E 5 (R1) [Ethnic Factors in the Acceptability of Foreign Clinical Data]: The study site is Pohnpei State, Federated States of Micronesia (FSM). Under US law and the Compact of Free Association between the US and FSM, this site is considered to be part of the US. There are no intrinsic (genetic or physiologic) or extrinsic (cultural or environmental) characteristics of the population that would influence the safety, efficacy, dosage or dose regiment of the drug. Children consume a diet largely of processed foods from the US mainland and the main pathogenic organism in the etiology of tooth decay has been shown to be *Streptococcus mutans*, as it is among children in the US proper. These children also use toothpastes produced in the US and regulated by FDA. In addition, this trial will be supervised by a regulatory monitor based in the US and familiar with US regulations.

# SCHEMATIC OF STUDY DESIGN



# 1. Key Roles

| Individuals: | |
|---|---|
| Principal Investigator: | Dr. Ohnmar Tut Department of Oral Health Sciences University of Washington, Seattle Email: Ohnmar@uw.edu |
| Sponsor/Investigator: | Peter Milgrom, DDS Member Advantage Silver Dental Arrest, LLC Email: drmilgrom@silverarrest.com |
| Medical Monitor | Johnny Hedson, MD<br>Pohnpei State Hospital<br>Pohnpei, FSM |
| Regulatory Monitors: | Douglas Bierer, PhD (primary) Douglas Bierer Consulting, LLC 7415 Graves Rd Cincinnati, OH 45243 William Cooley, PhD (secondary) Cooley Consulting, Inc. 531 Chisholm Trail Wyoming, OH 45215 |
| Site Director | Marcelle Gallen, BDS Chief of Dental Division Pohnpei State Department of Health Services Pohnpei, FSM |
| Institution and Locations: | Pohnpei State Department of Health Services Pohnpei, FSM |
| Biostatistician | Lloyd Mancl, PhD Research Associate Professor of Oral Health Sciences University of Washington Seattle, WA Email: Ilman@uw.edu |
| Coordination Center | Regional Clinical Dental Research Center<br>Institute of Translational Health Sciences<br>1959 NE Pacific St., Box 357480, Seattle, WA 98195<br>206-685-8132 / FAX: 206-685-9654 |

# 2. Introduction: Background Information and Scientific Rationale

# 2.1 Background Information

**Background:** Topical fluorides have been the mainstay in the prevention of dental caries for decades. There are abundant data on sodium fluoride's (NaF) ability to foster remineralization of tooth enamel (Gao et al., 2016). Dental NaF varnish preparations are the recommended vehicle for delivering topical NaF for dental caries prevention and arrest in young children under 6 years of age according to guidelines from the American Dental Association (ADA), the American Academy of Pediatrics, the American Academy of Pediatric Dentistry and the US Preventive Services Task Force (Weyant et al., 2013; Clark et al., 2014; American Academy of Pediatric Dentistry, 2013; Moyer VA 2014). In children, less than 6 years of age, at high risk for dental caries, the recommendation is application of NaF varnish every three months (Weyant et al., 2013). Fluoride varnishes have been shown safe in very young children (Milgrom et al., 2014).

However, topical fluorides alone are not enough to prevent tooth decay in high-risk populations. Caries researchers for some time have suggested strategies that combine topical antiseptic application to reduce or eliminate tooth surface colonization by cariogenic bacteria in addition to topical fluoride applications that primarily remineralize enamel (Milgrom et al 2009). Povidone iodine is an FDA-approved and widely used bactericidal antiseptic. For the oral flora, iodine has preferential activities against streptococcal species, pathogens implicated in the causation of dental caries (Tam et al., 2006; Furiga et al., 2008). Moreover, iodine's effectiveness may last as long as 6 months (Caufield et al., 1979).

Studies have examined the chemotherapeutic suppression of oral *Streptococcus mutans* (Sm) by povidone iodine (10%) in children with Severe Early Childhood Caries (S-ECC). In one study, the teeth of children two to six years of age were treated topically with povidone iodine (10%) or saline following dental treatment under general anesthesia for S-ECC (Zhan et al, 2006). Levels of Sm were significantly reduced up to three months in the povidone iodine group. A second study demonstrated suppression of Sm up to 90 days in children with S-ECC who received a single application of povidone iodine (10%) followed by a topical application of 1.23% acidulated phosphate fluoride foam after surgical elimination of active caries lesions (Berkowitz et al 2009).

Other studies have assessed the effect of povidone iodine (10%) on dental caries. A clinical study involving babies in Puerto Rico who were at high risk for S-ECC as they were all colonized by Sm and had decay-promoting feeding behaviors, demonstrated that povidone iodine (10%) applied bimonthly was successful in preventing the development of early tooth decay lesions in the maxillary primary incisors (Lopez et al., 2002). In a randomized clinical trial, povidone iodine (10%) applied bi-monthly significantly reduced the rate of recurrent dental decay at six months following treatment of children under general anesthesia for S-ECC (Amin et al., 2004).

Two cohort studies have tested the effect of combining these two anti-caries agents by sequentially applying povidone iodine (10%) followed 5% NaF varnish. The first study assessed the effect of protecting erupting 1<sup>st</sup> permanent molars from developing dental caries in children


five to six years old (Tut & Milgrom, 2010). The second studied the effect in the primary dentition of children 12 to 30 months (Milgrom, Tut & Mancl, 2011). They demonstrated that treatment with povidone iodine reduced the rate of new decay significantly over the standard of care alone. Yet, to date, such combination products have not been brought to the market. Advantage Anti-Caries Varnish was developed to combine the antiseptic povidone iodine and sodium fluoride varnish into a single product for ease of application, particularly in high caries risk, preschool age children.

A phase 1 study of the safety of the new varnish was conducted in 12 healthy children with an average age of 47.6 months (WIRB PRO NUM: 20160539). No child evidenced any intra oral erythema or secondary changes as a consequence of the varnish application either immediately or within 24-48 hours post application. Neither were there any adverse effects. The FDA has reviewed the previous safety work and this protocol and issued IND 128835 for this work.

A phase 1 study (Lin, Rothen & Milgrom, 2018) was carried out to characterize the kinetics of iodine and fluoride following topical application of the PVP-I and NaF anti-caries varnish in healthy adults (WIRB PRO NUM: 20161181). Sixteen subjects (23 to 57 years) participated in a pharmacokinetics study following the application 0.4 mL of a varnish containing 10% (w/v) PVP-I and 5% (w/v) NaF. Serum and urine samples were collected at various time points over 24 hours following application of varnish. Iodine and fluoride concentrations were analyzed, and for each time point baseline concentrations were subtracted from observed values. Following varnish application, 2 of 16 participants had nearly undetectable baseline-corrected iodine and fluoride levels, suggesting minimal absorption, lack of release iodine and fluoride from the varnish, or inconsistent dosing. The average peak concentrations were 57 ± 33 ng/mL iodine and  $60 \pm 34$  ng/mL (0.060  $\pm$  0.034 ppm) fluoride and occurred within 3 hr of application. The average elimination half-life was 5.5 ± 1.4 hr and 3.1 ± 1.6 hr for iodine and fluoride. respectively. Renal clearance of iodine and fluoride were similar to literature values. No adverse events related to the study varnish were observed by the investigative team or reported by the participants. In this study, serum fluoride and iodine transiently increased, but were within normal range 24 hr after application of the varnish. This study has shown that the combination of PVP-I and NaF in a proposed anti-caries varnish was well tolerated.

Phase 2 Study in FSM. A single center randomized, double-blind, active-controlled, parallel-group trial to assess efficacy of the Advantage Anti-Caries Varnish (10% PVP-I, 5.0% NaF) was conducted in Pohnpei FSM to determine if it is superior to a varnish containing only 5% NaF in the prevention of new caries lesions (COM-FSM IRB Protocol #2017-18-05; WIRB PRO NUM: 20170090). The study population was healthy children 48 to 84-months-old enrolled in 10 Early Childhood Education centers. There were 299 consents in a school population of 377 children. A study assistant collected healthy history information. Fifteen children were excluded and 284 were randomized (1:1 allocation). Two hundred seventy-three children were analyzed in year 1 and 262 children were analyzed in year 2. The dental varnish contained 10% PVP-I and 5.0% NaF. The comparator contained only NaF. Varnishes were applied once every 3 months during two years. The primary outcome was the surface-level primary molar caries increment (d<sub>2-4</sub>mfs) at two-years. Baseline to Year 1 and Year 2, caries increments were compared between conditions using log-linear regression adjusting for age, sex and baseline caries and whether the tooth was sound (free of caries lesions) at baseline. At year 1, the caries increment for primary molars sound at baseline was 0.9 surfaces (SD 1.5) for the test varnish


versus 1.8 (SD 2.2) for the varnish with fluoride alone (adjusted RR=0.50; 95% CI: 0.31 to 0.81; P = .005). At year 2, the caries increment for primary molars sound at baseline was 2.3 surfaces (SD 2.8) for the test varnish versus 3.2 (SD 2.6) for the varnish with fluoride alone (adjusted RR=0.74; 95% CI: 0.52 to 1.03; P = .073). Teeth that were already cavitated at baseline did not show a secondary preventive effect. There were no harms. Results confirm the results of an earlier cohort study suggesting a dental varnish containing PVP-I and NaF is effective in the primary prevention of cavities in the primary dentition.

The basic dental varnish formula was previously cleared by the FDA as a medical device and is currently on the market. To our knowledge there have been no adverse event reports on this varnish and it has never been withdrawn from the market. Povidone iodine is widely used in children in medicine. It has been used for intraoral application for many years without problems. Dental NaF varnish and povidone iodine have been applied sequentially at the same patient visit by clinicians for some time and two cohort studies have been published with no reports of harms. Similarly, the recently completed Phase 2 trial reported no harms.

# 2.2 Potential Risks and Benefits

#### 2.2.1 Potential Risks

None of the proposed methods pose any serious risks to the study subjects.

The FDA approves the topical use of 10% PVPI to the skin of children.

Risks from povidone iodine include rash and swelling at the site of application. lodine can cause thyroid gland problems, but this is rare and is very unlikely at the amount used in this study.

The recent phase 2 trial demonstrated no harms.

#### 2.2.2 Known Potential Benefits

There are direct benefits to the human subjects participating in this proposal. These include the early detection of caries, its timely management and the possibility of its prevention.

# 3. Objectives

#### 3.1 Study Objectives

Primary Objective:

To determine if Advantage Anti-Caries Varnish (test varnish) is superior to an active control varnish (5% NaF) in the prevention of caries lesions in the primary dentition (Severe-Early Childhood Caries). Specifically, prevention of caries lesions in primary teeth that either are sound, have only d<sub>1</sub> (white spots) lesions or unerupted at baseline.

Secondary objectives:

To document the safety of the test varnish.

# 3.2 Study Outcome Measures

#### 3.2.1 Primary Outcome Measures

- New surface-level dental caries lesions at 24 months post baseline
- Presence/Absence of any new dental caries lesions (d<sub>2-4</sub>mfs) at 12 months post baseline

#### 3.2.2 Secondary Outcome Measures

Adverse event occurrence

#### 4. Study Design

This is a single center randomized, double-blind, placebo-controlled, parallel-group trial.

# 4.1 Rationale for Study Design

The completed phase 2 study demonstrated a preventive effect on primary teeth that were sound (not cavitated) at baseline but the study was not specifically designed to test the primary prevention efficacy. The hypothesis in this second phase 2 study is that the test varnish will be superior to the active control varnish for primary prevention of S-ECC. There will be no difference in the frequency of adverse events.

# 4.2 Rationale for Dosage

The treatment group will be exposed at baseline and once every three to four months after baseline for a maximum period of 24 months. The control group will be exposed to the control varnish in the same manner. The decision for dosing every three to four months with the test varnish was based on earlier work (Berkowitz, Koo et al. 2009) and the AAPD Standard of Care for children at high risk for dental caries.

# 5. Study Enrollment and Withdrawal

#### 5.1 Subject Numbers

254 subjects will be enrolled. Half will be randomized to each arm.

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

# 5.2 Subject Inclusion Criteria

- 1. The subject's parent or legal guardian must provide signed and dated informed consent (parent permission form).
- 2. The subject's parent or legal guardian of the subject must be willing and able to comply with study requirements.
- 3. The subject is a 6 to 24 months at the time of enrollment.
- 4. The subject must be in good general health as evidenced by parent report.
- 5. The subject will have at least 1 erupted tooth that is either sound or has only a d<sub>1</sub> (white spots) lesion.

#### 5.3 Subject Exclusion Criteria

A subject who meets any of the following criteria will be excluded from participation in this study:

- 1. Previous treatment with fluoride varnish
- 2. Known allergy to iodine
- 3. Diagnosis of thyroid disease
- 4. Chronic, prophylactic use of antibiotics
- 5. Treatment with another investigational drug or intervention within 30 days preceding the Baseline Visit.
- 6. Visible cavities (d<sub>2-4</sub>)

- 7. Presence of intraoral pathology that would make assessment of post treatment soft tissue ulcerations or inflammation impossible (child could be enrolled if problem is treated and lesions cleared)
- 8. Parent anticipates the child will move from Pohnpei during the next 2 years.

In the event of unique circumstances permitting waiver of any of the above eligibility criteria, documentation of such a waiver must be generated by the Principal Investigator prior to randomization into the study. Enrollment of an otherwise ineligible subject into the study without prior approval of a waiver will be considered a protocol violation.

# 5.4 Discussion of Subject Characteristics

The study population is high risk for Severe-Early Childhood Caries (any dental caries in the primary dentition before the age of 5) because of their poverty status and lack of access to fluoridated water. The subject population will consist of children who are 10 to 20 months of age at the time of enrollment. The study site is Pohnpei State, Federated States of Micronesia (FSM). Under US law and the Compact of Free Association between the US and FSM, this site is considered to be part of the US. There are no intrinsic (genetic or physiologic) or extrinsic (cultural or environmental) characteristics of the population that would influence the safety, efficacy, dosage or dose regiment of the drug. Children consume a diet largely of processed foods from the US mainland and the main pathogenic organism in the etiology of tooth decay has been shown to be *Streptococcus mutans*, as it is among children in the US proper. These children also use toothpastes produced in the US and regulated by FDA. In addition, this trial will be supervised by a regulatory monitor based in the US and familiar with US regulations. The consent documents will be in English and Pohnpeian.

#### 5.5 Strategies for Recruitment and Retention

Children attending Maternal and Child Health (MCH) Immunization and Well Child programs in Pohnpei State will be enrolled. In 2019 there were 6 MCH centers and a Community Health Center enrolling 597 children. In this age range there will be at least 500 children available to recruit. Assuming a consent rate of 80% (allowing for a few children with cavities and some moving off island), we should be able to recruit 254 children in less than 3 months. Based on the recently completed phase 2 trial and our previous work in Micronesian schools in the US affiliated states we expect nearly every parent to consent and thus for us to enroll the entire sample within two months (Milgrom et al., 2009; Tut et al., 2010; Milgrom et al., 2011).

The parent (or legal guardian) of the potential subject will be approached by a bilingual study assistant who will confirm eligibility of the subject. The proposed study will be explained. Written informed consent will be obtained. The child will be screened for presence of dental cavities. If the child is cavity free and meets all the inclusion criteria, he/she will be enrolled in the study and randomized according to the randomization list created by the study biostatistician.

The Micronesian islands are quite isolated and children do not move from the islands readily. In the recently completed phase 2 trial, less than 10% of children were lost to follow-up after two years. We have conducted two prospective cohort studies with a similar population in the islands. The one-year attrition rate was 1/172 (less than 1%) in one study and no child was lost to follow-up in the other study (Tut & Milgrom, 2010; Milgrom, Tut & Mancl, 2011). Families whose children complete the first treatment visit will receive a \$20 gift card as an incentive and then receive an additional \$20 gift card at each 3-month treatment visit. Families whose children complete a year in the study will receive a \$30 gift card at the Year 1 dental examination; families whose children complete two years in the study will receive a study t-shirt at enrolment. All child participants will receive a small tube of fluoridated toothpaste and an appropriately sized toothbrush at treatment visits. The incentive levels were determined in consultation with the Pohnpei State Department of Health and Social Services.

# 5.6 Treatment Assignment Procedures

#### 5.6.1 Subject Identification Numbers

Participants will be randomly assigned to one of the two inventions with a 1:1 allocation as per a computer-generated randomization schedule with stratification by MCH center (Nett, Kolonia, Kitti and Sokehs if needed) and with randomly permuted blocks of sizes 2 and 4. Multiple children within the same family unit will be randomized independently. Stratification and blocking will ensure the two interventions are equally balanced within MCH center and randomly permuted blocks sizes will ensure concealment.

#### 5.6.2 Randomization Procedures

The study biostatistician will create the randomization lists using the "sample" function of the R statistical software (Version 3.3.0; The R Foundation for Statistical Computing, 2016).

The biostatistician will generate treatment assignment lists for each MCH center. Treatments will be blinded and coded drug A or B. In each treatment application a second staff member will verify on site that the child received the correct coded treatment.

#### 5.7 Masking Procedures

All study personnel except for designated personnel in the data center will be blinded to the participant treatment assignment. In order to maintain blinding and eliminate examiner bias, the staff member applying these varnishes will not perform the caries scoring exams.

#### 5.8 Reasons for Withdrawal

Subjects' parents or legal guardians will be advised in the written consent that they have the right to withdraw from the study at any time without prejudice, and may be withdrawn at the Principal Investigator's discretion at any time.

A subject may be withdrawn from the study for the following reasons:

Examples of non-adverse-event related reasons for withdrawal

- 1. Withdrawal of consent by parent/guardian
- 2. Principal Investigator-initiated withdrawal
- 3. Request of primary care physician
- 4. Failure to meet entry criteria (either newly developed or not previously recognized)
- 5. Lost to follow-up/failure to return
- 6. Early termination of study

Examples of adverse event-related reasons for withdrawal

- 1. New illness that in the opinion of the Principal Investigator warrants withdrawal
- 2. Death
- 3. Other adverse event

#### 5.8.1 Handling of Withdrawals

In the event of voluntary withdrawal from the study, a Premature Withdrawal (PW) Visit will be conducted if possible to obtain a final caries exam and ensure that appropriate care under medical supervision is provided until the symptoms of any AE resolve or the subject's condition becomes stable or deemed chronic.

Reasonable effort should be made to contact any subject lost to follow up during the course of the study in order to complete study-related assessments and collect safety data.

Subjects who are withdrawn from the study will not be replaced.

# 5.9 Termination of Study

The study may be discontinued at the discretion of the Sponsor or the Principal Investigator if there is sufficient reasonable cause.

Circumstances that may warrant termination include, but are not limited to:

#### Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention

Protocol # 2019-10-19


- Determination of unexpected, significant, or unacceptable risk to subjects.
- · Insufficient rate of subject accrual.
- Insufficient adherence to protocol requirements.
- Data which are not sufficiently complete and/or evaluable.

Written notification, documenting the reason for study termination, will be provided to the Principal Investigator and regulatory authorities. In the event of early termination of the study, all subjects will be seen for a final visit for safety purposes. The study site will notify the Western IRB and the Pohnpei State Department of Health and Social Services of the study termination and provide the reason(s).

# 6. Investigational Product

# 6.1 Investigational Product Description

# 6.1.1 Acquisition

Test and control varnishes will be obtained from Cascade Custom Chemistry, Eugene, OR

#### 6.1.2 Formulation, Packaging, and Labeling

Advantage Anti-Caries Varnish. The active ingredients are 10% (w/v) Povidone lodine CAS RN 25655-41-8 and 5% (w/v) Sodium Fluoride CAS RN 7681-49-4 in Ethanol 200 Proof. The formulation of the dosage form includes 10% Nt-2 Premium Shellac, 1% sodium phosphate, dibasic anhydrous, 0.5% ammonium phosphate, monobasic, and 1% caramel cream flavor (Bell 29.26303) as inactive ingredients. One and two-year shelf life of the varnish has been established according to Guidance for Industry Q1A(R2) Stability Testing of New Drug Substances and Products (Revision 2, November 2003).

The active control varnish will be the same varnish without iodine with an appropriate FDA approved food dye added to match the color of the test agent. There will be no other differences in the treatment and control varnishes.

The varnishes will be packaged in 12 mL multi use bottles with the following labeling.

#### Advantage Anti Cavity Varnish or Control Varnish

- Apply as per protocol
- For Investigational Use Only
- Drug Code A or B

• Contact: Dr. Peter Milgrom, +1206-251-6831 (24 hours)

# 6.1.3 Product Storage and Stability

All investigational products will be kept in a secure, safe area under recommended storage conditions with access limited in the study office. Expiration or use-by dates, as applicable, for all products will be documented by staff.

# 6.2 Dosage, Preparation and Administration of Study Investigational Products

## Advantage Anti-Cavity Varnish and Control Varnish

A maximum of 0.2 mL will be applied to the teeth with a dental brush. Test or control varnish will be applied topically 4 times per year following enrollment and at each 3 to 4-month intervals.

The specific procedure is as follows. The varnish multi-use vial is shaken for 1 minute before dispensing. The varnish will be dispensed into the well of the disposable plastic dappen dish. One drop will be dispensed for every five teeth to be treated, up to a maximum of 4 drops if all 20 primary teeth are present. Teeth will be dried with cotton gauze prior to application. Varnishes will be applied to the teeth with a dental microbrush.

### 6.3 Accountability Procedures for the Investigational Product(s)

The Principal Investigator (Tut) and Site Director (Gallen) must maintain accurate records (including dates) of all supplies received from Advantage. All remaining drug will be returned to the sponsor for disposal and documented on the Drug Disposal Log by the Sponsor or Principal Investigator.

# 6.4 Assessment of Subject Compliance with Investigational Product

As the test and control drugs will be administered by the study personnel, it is not anticipated that subject compliance with treatment will be an issue. In the event a dose is missed; the missed dose will be captured as a protocol deviation and documented in the source documents.

#### 6.5 Coding/Emergency Treatment Disclosure

The Principal Investigator will be given a sealed envelope containing the randomized treatment assignment code for each subject to be opened only in the event of a medical emergency.

Neither premature withdrawal from the study nor most clinical emergencies necessitate disclosure of treatment assignment. Most emergency situations can be handled by withdrawing study treatment without disclosure of treatment assignment. However, in rare circumstances under which knowledge of the drug assignment is necessary for the treatment of a serious adverse event, the Principal Investigator (Tut) must discuss the situation with the Site Director (Gallen) and Dr. Milgrom, if circumstances permit, before deciding whether or not to disclose treatment assignment. If disclosure of individual treatment assignment is undertaken, it must be made by the Principal Investigator responsible for the care of the involved subject in consultation with the Medical Monitor. The subject will be withdrawn from further exposure to study drug.

Emergency treatment is a reportable event, requiring notification to the Principal Investigator and Sponsor within 24 hours when the staff is aware of the event. The assigned treatment must not be revealed to other study staff or to individuals who are not involved directly in the clinical care of the subject, unless disclosure to the individual is critical to the care of the subject.

#### 6.6 Concomitant Medications/Treatments

Subjects may not be receiving treatment with another investigational drug within 30 days preceding the baseline visit and throughout participation in this study.

Chronic prophylactic use of antibiotics at enrollment is an exclusion criterion; however, if during the course of the study, the subject's PCP prescribes antibiotics (e.g., for treatment of otitis media) the subject can remain in the study. At each varnish application, the study staff will question the parent about antibiotic use as part of capturing AEs and this will be recorded on the AE form.

Concomitant medication use, including all prescription and over-the-counter medications, will be recorded commencing with the screening visit and at each visit through completion of the study.

Fluoridated toothpaste will be provided under this protocol to all subjects. Parents will be given a handout explaining how much toothpaste to use. At each follow-up, the parent will be asked about whether the child is using the fluoride toothpaste. The parent will be asked to estimate about how many times per week, in a typical week, that their child is using the fluoride toothpaste (e.g., every day, more than half the days, less than half the days, never).

# 7. Study Schedule/Procedures and Evaluations

#### 7.1 Subject recruitment procedures:

 The study assistant will contact the parent/caregiver through the MCH Immunization or Well Baby program or at home. This individual will explain the study and obtain

- informed consent. The focus will be on Nett, Kolonia, and Kitti districts. Sokehs will be included if necessary.
- The informed consent packet will carry a pre-assigned subject number. If a parent does not consent, the reason will be recorded and the study number will not be used.
- The study assistant will verify that the subject meets the inclusion and exclusion criteria, including age. The study assistant will calculate from the birth date that the subject is at least 40 6 months of age exactly and no more than 20 24 months and 0 days.
- The study assistant will record the subject's age and sex and medical history based on parent/guardian report.
- The study assistant will record concomitant prescription medication and over-the-counter medication use over the past 90 days.
- A trained and calibrated study dental assistant will conduct the baseline dental screening for cavities, chart the number of fully and partially erupted teeth, and any abnormal intraoral soft tissue findings.
- If the child meets the Subject Inclusion Criteria, the child will be enrolled for the study and entered into the randomization list created by the Study Biostatistician for treatment.

#### 7.2 Baseline Visit

- The visit will be at a center or at the study office.
- At the baseline visit, the Project Site Manager will check the randomization list and the drugs, which will be color-coded, and a trained study dental assistant will apply the first treatment to the subject according to the treatment code assigned by the statistician.
- A toothbrush and a small tube of fluoride toothpaste will be dispensed to the parent/caregiver along with a handout explaining how much toothpaste to use.
- 24-48 hours later, a trained study dental assistant will see the child again and conduct a soft tissue exam, and complete the safety questionnaire.

#### 7.3 Visits 2-8 Treatment Visit

- The visit will either be at a MCH/CHC Center or the study office.
- A trained study dental assistant will review and record adverse events (AEs) and concomitant prescription and over-the-counter medications.
- Fluoride toothpaste use will be collected from the parent/caregiver and recorded by a trained study dental assistant.
- A trained and calibrated examiner will conduct the dental caries exam at Visit 5 (Year
   1).
- A trained study dental assistant under the direction of the Project Site Manager, who will consult the participant list and randomization, will apply the assigned treatment.

- A toothbrush and a small tube of fluoride toothpaste will be dispensed to the parent/caregiver along with a handout explaining how much toothpaste to use.
- 24-48 hours later, a trained study dental assistant will telephone the parent and
  assess any adverse or serious adverse event and complete the safety questionnaire.
  If the parent cannot be contacted the assistant will make a home visit or arrange for
  the child to be brought to study office. If there is an apparent adverse or serious
  adverse event, the child will be seen in person by study staff. see the child again,
  conduct a soft tissue exam, and complete the safety questionnaire.

#### 7.4 Visit 9 Year 2 Exam Visit

- The visit will either be at a MCH/CHC Center or the study office.
- A trained study dental assistant will review and record adverse events (AEs) and concomitant prescription and over-the-counter medications.
- Fluoride toothpaste use will be collected from the parent/caregiver and recorded by a trained study dental assistant.
- A trained and calibrated examiner will conduct the dental caries and oral exam (Year 2).

#### 7.5 Premature Withdrawal

In the event of premature withdrawal from the study, the Premature Withdrawal (PW) visit procedures and evaluations should be completed whether or not the decision to withdraw is determined at a routine or unscheduled visit. If it is determined via telephone contact that a premature withdrawal will occur, the parent/guardian should be asked to bring the child in for a PW visit.

Activities to be completed include:

- The Examiner will conduct the Oral Soft Tissue exam
- The Examiner will conduct the caries exam
- The assistant will record concomitant medication use.
- The assistant will review and record AEs and record on the AE Follow-Up Log the status
  of adverse events that are unresolved at the time of the premature withdrawal visit.

Premature withdrawal (including reports of subjects who are lost to follow up) should be reported to the Site Director within 24 hours of the site's knowledge of the event.

#### 7.6 Unscheduled Visit

An unscheduled visit may be performed at any time during the study at the subject's request or as deemed necessary by the Principal Investigator. The date and reason for the unscheduled visit will be recorded in the subject's source documentation.

Activities to be completed include:

- The Examiner will conduct the Oral Soft Tissue exam
- The Examiner will conduct the caries exam
- The assistant will record concomitant medication use.
- The assistant will review and record AEs and record on the AE Follow-Up Log the status
  of adverse events that are unresolved at the time of the unscheduled visit.

### 8. Assessments

# 8.1 Primary and Secondary Outcome Variables

Primary Outcome Variable

- Surface-level dental caries lesions (d<sub>24</sub>mfs) at 24 months post baseline
- Presence/Absence of dental caries lesions (d<sub>2-4</sub>mfs >0) at 12 months post baseline

Secondary Outcome Variable: Adverse Events

# 8.2 Efficacy Assessments

#### 8.2.1 Caries Examination

Two examiners will be trained and calibrated according to National Institute of Dental and Craniofacial Research Early Childhood Caries Collaborative criteria, which are based on the World Health Organization caries classification system. The children will be visually examined using a mouth mirror and artificial light. No explorers will be used. Training and calibration will be done prior to dental exams at year 1 and year 2. At each timepoint, six subjects will be used for training and 14 subjects will be used to evaluate examiner agreement.

#### 8.3 Safety Assessments

Adverse events, including frequency and severity, and perceived relationship to the investigational product, will be compared between the treatment groups.

# 8.3.1. General Health (Medical History and Physical Examination)

The subject's general health status at enrollment will be assessed by medical history using the parent or legal guardian as the informant.

The Study Site Manager will rule out a history of thyroid disease and iodine allergy.

All concomitant medications taken by the subject will be recorded at the time of consent and updated at each follow-up study visit (all prescription and over-the-counter medications taken within the past three months).

#### 9. Assessment of Safety

# 9.1 Specification of Safety Parameters

Adverse events

# 9.2 Methods and Timing for Assessing, Recording, and Analyzing Safety Parameters

Adverse events will be recorded at each 24-48 hour in person or telephone check. At each treatment visit, the parent will be questioned about any changes in the child's health and AEs noted.

Adverse events will be reviewed on a quarterly basis by the Medical Monitor (Hedson); serious adverse events and other protocol-specified reportable events will be assessed in real time by the Principal Investigator (Tut) and Site Director (Gallen).

#### 9.3 Adverse Events

An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with any use of a drug, whether or not related to the drug. An adverse event can arise from any use of the drug (e.g., off-label use, use in combination with another drug) and from any route of administration, formulation, or dose. This excludes minor fluctuations in signs or symptoms of the disease under study, but does include significant worsening of the disease. It also includes any apparently unrelated illness and any accident that occurs during participation in the study.

Some examples of adverse events are:

- Development of an illness during the study.
- Development of symptoms which may or may not be related to the use of a concomitant medication or investigational product.

All adverse events, whether observed by the Principal Investigator, elicited from or volunteered by the subject or parent/guardian, should be recorded on a study Adverse Event Form and in the Adverse Event Log. This reporting will include a brief description of the

event, the date of onset, the date of resolution, the duration and type of event, the severity, contributing factors, and any action taken with respect to the investigational product.

AEs occurring after informed consent is obtained but prior to randomization will be recorded as medical history, unless possibly related to a study procedure, in which case they will be recorded as adverse events in the case report form. New adverse events will be captured and reported on the AE log until 30 days following the last treatment or premature withdrawal, whichever comes first.

#### 9.4 Expected Adverse Reactions

Risks from povidone iodine include rash and swelling at the site of application. Iodine can cause thyroid gland problems.

#### 9.5 Serious Adverse Events

A serious adverse drug event is defined as any adverse event that results in any of the following outcomes:

- death
- a life-threatening adverse event
- inpatient hospitalization or prolongation of existing hospitalization
- a persistent or significant incapacity; or substantial disruption of the ability to conduct normal life functions
- [a congenital anomaly/birth defect noted as not applicable in this population]

An important medical event that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, the event may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include (but are not limited to) allergic bronchospasm requiring intensive treatment in an emergency room or at home, or blood dyscrasias or convulsions that do not result in inpatient hospitalization.

This category also includes any event the Principal Investigator judges to be serious or that would suggest a significant hazard, contraindication, side effect or precaution. Any adverse event or suspected adverse reaction is considered "life threatening" if, in the view of either the Principal Investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

Reports of serious adverse events require immediate notification (within 24 hours of the site's awareness) to the Principal Investigator and Sponsor whether or not the Study Site Coordinator believes that the event is related to investigational product or is expected.

#### 9.5.1 Unanticipated Problems

The Principal Investigator must conform to the adverse event reporting timelines, formats and requirements of the various entities to which she is responsible, but at a minimum those events that must be reported are those that are:

- · related to study participation,
- unexpected, and
- serious or involve risks to subjects or others

#### 9.5.2 Procedures to be Followed in the Event of Abnormal Clinical Findings

At each child 24-48-hour follow-up, study staff will assess adverse events by assessment of parent report and clinical features if the child is seen in person and parent questionnaire.

An unscheduled visit may be performed at any time during the study as deemed necessary by the Principal Investigator. The Site Director will inform the subject's parent/guardian when medical care is needed for adverse events of which the Principal Investigator becomes aware (e.g., illness) and may refer the subject back to the PCP for further work-up. The Principal Investigator may determine that the subject should be withdrawn from the study treatment.

# 9.6 Reporting Procedures

#### 9.6.1 Reportable Events

The following incidents will be considered reportable events and will be reported to the Principal Investigator within 24 hours of the site's awareness of the event.

- Serious Adverse Event
- Emergency Treatment Disclosure
- Post-Treatment Adverse Events, including
  - Nausea
  - Not eating
  - Vomiting
  - Difficulty swallowing or breathing
  - Swelling around the lips or skin on the face
  - o Itchiness around the lips or skin of the face
  - Hives or rash

# 9.6.2 Serious Adverse Events

Within 24 hours of the site's awareness of the serious adverse event (SAE), the site will report the SAE to the Principal Investigator and provide subject identification and a brief description of the event, including the Medical Monitor's

assessment of causality (unrelated, possible, probable, definite) related to the study drug.

Within 24 hours of the telephone report, the site will complete the AE form and update the AE log to ensure that the concomitant prescription medication information is current, and enter the SAE report. This report will include: documentation that serious adverse event criteria have been met; a detailed description of the event and other relevant information; the current status of the experience; if the subject has died, the date of death and autopsy report, if available; and the Medical Monitor's current opinion of the relationship between the event and the investigational treatment.

# 9.6.3 Adverse Event Causality Definitions

For each adverse event, the relationship to the study drug (Medical Monitor's attribution of causality) must be recorded as one of the following on the Adverse Event Log:

| TERM | DEFINITION | CLARIFICATION |
|---|---|---|
| Unrelated | No possible relationship | The temporal relationship between drug exposure and the adverse event onset/course is unreasonable or incompatible, or a causal relationship to study drug is implausible. |
| | Not reasonably related, although a causal relationship cannot be ruled out | While the temporal relationship between drug exposure and the adverse event onset/course does not preclude causality, there is a clear alternate cause that is more likely to have caused the adverse event than the study drug. |
| Possible | Causal relationship is uncertain | The temporal relationship between drug exposure and the adverse event onset/course is reasonable or unknown, dechallenge or rechallenge information is either unknown or equivocal, and while other potential causes may not exist, a causal relationship to the study drug does not appear probable. |
| Probable | High degree of certainty for causal relationship | The temporal relationship between drug exposure and the adverse event onset/course is reasonable. There is a clinically compatible response to dechallenge (rechallenge is not required), and other causes have been eliminated or are unlikely. |
| Definite | Causal relationship is certain | The temporal relationship between drug exposure and the adverse event onset/course |


| TERM | DEFINITION | CLARIFICATION |
|------|------------|-------------------------------------------------|
| | | is reasonable, there is a clinically compatible |
| | | response to dechallenge, other causes have |
| | | been eliminated, and the event must be |
| | | definitive pharmacologically or |
| | | phenomenologically, using a satisfactory |
| | | rechallenge procedure if necessary. |

# 9.6.4 Adverse Event Severity Definitions

The severity of each adverse event must be recorded as one of the following on the Adverse Event Log:

MILD No limitation of usual activities
MODERATE Some limitation of usual activities
SEVERE Inability to carry out usual activities

# 9.7 Responsibilities of Investigator/Sponsor for Reporting SAEs

Serious adverse events occurring after informed consent is obtained but prior to randomization will be recorded as medical history, unless possibly related to a study procedure, in which case they will be reported as SAEs to the Medical Monitor within 24 hours of the site's awareness.

# 9.7.1 Regulatory Reporting for Studies Conducted Under an IND

The Principal Investigator will comply with the Micronesian and Western IRB regulations regarding the reporting of adverse events.

The Sponsor will report events that are <u>serious</u>, <u>unexpected</u> and that are <u>associated</u> with the study drug (SUSAR) to the Food and Drug Administration (FDA) within the required timelines as specified in 21 CFR Part 312.32; fatal and life-threatening events within 7 calendar days (by phone or fax) and all other SAEs in writing within 15 calendar days. All serious events designated as "not associated" with study product(s) will be reported to the FDA at least annually in a summary format.

#### 9.7.2 Other Unanticipated Problems

Unanticipated problems are those involving risks to subjects or others and include any incident, experience, or outcome that meets **all** of the following criteria:

- Unexpected (in terms of nature, severity, or frequency) given (a) the research procedures that are described in the protocol-related documents, such as the WCG IRB-approved research protocol; and (b) the characteristics of the subject population being studied;
- Related or possibly related to participation in the research (possibly related means there is a reasonable possibility that the incident, experience, or outcome may have been caused by the procedures involved in the research); and
- Suggests that the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized.

An incident, experience, or outcome that meets any of the three criteria above generally will warrant consideration of substantive changes or corrective actions in order to protect the safety, welfare, or rights of subjects or others.

Unanticipated problems noted by the site will be recorded and reported to the Principal Investigator within 24 hours of the site's awareness and to the Micronesian and WCG IRB per local reporting requirements.

# 9.8 Type and Duration of Follow-up of Subjects after Adverse Events

All adverse events will be followed until resolution or an appropriate endpoint is reached (e.g., the Medical Monitor attributes the adverse event to a cause other than the study drug or assesses it to be chronic or stable).

# 9.9 Halting Rules

Adverse events, particularly serious adverse events such as deaths and hospitalizations, will be carefully considered by the Sponsor. If necessary, the Sponsor will halt the study.

#### 10. Site Monitoring

#### 10.1 Clinical Site Monitoring

To ensure compliance with Good Clinical Practice (GCP) and other applicable regulatory requirements, the Regulatory Monitor (Bierer) is responsible for monitoring to ensure the site is conducting the study according to the protocol, Standard Operating Procedures (SOPs), and other written instructions and regulatory guidelines. Monitoring visits by a Regulatory Monitor will be arranged in advance, at a mutually-acceptable time, with site personnel.

The site personnel must allow sufficient time for the Regulatory Monitor to review CRFs and relevant source documents, including access to electronic medical records, and address data queries.

The Investigators should be available to answer questions or resolve data clarifications. The monitoring plan will include written procedures for periodic and closeout monitoring visit activities, documentation and communication of visit findings, and maintenance of the record of on-site visits. The monitoring plan will serve as a guide to ensure standardization of study-specific procedures for the Regulatory Monitor who is responsible for ongoing quality review.

# 10.2 Regulatory Inspections

During the course of the study and after it has been completed, it is possible that one or more study site visits will be undertaken by authorized representatives of the Sponsor, WCG IRB, or regulatory agencies, such as the Food and Drug Administration (FDA). These audits may take place at any time during or after the study and are based on the local regulations, as well as ICH guidelines.

The purpose of the audit is to determine whether or not the study is being, or has been, conducted and monitored in compliance with the protocol as well as recognized GCP guidelines and regulations. These audits will also increase the likelihood that the study data and all other study documentation can withstand a subsequent regulatory authority inspection.

If such audits are to occur, they will be arranged for a reasonable and agreed-upon time.

#### 11. Statistical Considerations

# 11.1 Study Hypotheses

The hypothesis is that the Advantage Anti-Caries Varnish (test varnish) is superior to an active control varnish (5% NaF, no PVP-I) in the prevention of caries lesions in the primary dentition (Severe-Early Childhood Caries), and there will be no difference in the frequency of adverse events. Specifically, prevention of caries lesion in primary teeth that either are sound, have only d<sub>1</sub> (white spots) lesions or unerupted at baseline.

#### 11.2 Sample Size Considerations

The study aims to show differences in the net caries increment ( $d_{2-4}$ mfs) at 2 years post baseline application (Broadbent & Thomas, 2015) and any new caries at 1 year post baseline. Assuming a coefficient of variation of 85% in the caries increment and a 35% reduction in caries increment at 2 years (equivalent to an effect size of 0.49), 106 children per group will be required for 90% power using a 0.025 significance level. With 106 children per group the power is 80% to show a 38% reduction in any new caries at 1 year using a 0.025 significance level assuming 55% caries in the control group. The effect sizes were based on the findings from our prior study on the test varnish involving 4-6 year-old children


and our study on topical iodine and fluoride varnish effectiveness involving 12-30 month-old children (Milgrom et al 2011). The sample size was inflated 20% to 127 per group to account for loss to follow-up, particularly for moving off island. The follow-up rate in our prior study in this population was >90% after two years.

# 11.3 Statistical Analysis Plan

### 11.3.1 Primary Statistical Analysis.

The primary analysis will be conducted in accordance with the intention-to-treat principle; and if needed, multiple imputation procedures will be used to account for missing caries information (Schafer, 1997). For the primary outcome at year 2, incremental dental caries based on d<sub>2-4</sub>mfs, the unit of analysis will be the child and the net dental caries increment will be compared between the two interventions at 2 years post baseline using a two-sample t test assuming unequal variances. The primary comparison will be based on all primary teeth and surfaces, and additional comparisons will be based on sound surfaces, surfaces with d<sub>1</sub> (white spots) or unerupted surfaces of primary teeth at baseline. This approach assumes the distribution of dental caries increment is approximately symmetrical, which is often true in high-risk caries populations. In the case of non-symmetry, log-linear regression using robust standard errors, which can accommodate count outcomes with a skewed distribution, will be used to compare the caries rates between the two interventions (Hardin & Hilbe, 2013), Log-regression analysis will use the tooth as the unit of analysis and be based on all teeth, but include an indicator for whether a tooth is sound, only has d<sub>1</sub> (white spots) lesions or unerupted at baseline, an interaction between this tooth indictor and intervention arm to allow for separate estimates and tests of the intervention effect based on the status of the tooth at baseline. Covariate-adjusted linear or log-linear regression models using robust standard errors will be used to compare dental caries increment, adjusting for baseline dental caries, stratification variables (MCH center), gender and age of the participant (Hardin & Hilbe, 2013). The log of the number of surfaces at risk will be included as an offset in the log-linear regression models.

Similar comparisons between the two intervention arms will be performed for the present or absence of any new dental caries  $d_{2-4}$ mfs >0) one-year post baseline. Unadjusted comparisons between the two intervention arms will done using the chi-square test and the child as the unit of analysis, and log-binomial regression with the tooth as the unit analysis will be used to compute adjusted relative risks and perform comparisons between the two intervention arms adjusting for baseline dental caries, stratification variables (MCH center), gender and age of the participant (Hardin & Hilbe, 2013).

If needed, pre-protocol analyses will be performed based on the number of varnish applications the child received. In our prior Phase 2 trial, children received all varnish applications per the protocol, or at least until the child was lost to follow-up. The proposed log-linear and log-binomial regression methods will be used to assess whether adjusting for toothpaste use affects the comparison between the two interventions and to test for effect

modification of an intervention effect by toothpaste use. Toothpaste use will be summarized for two time periods, between baseline and year 1 between year 1 and year 2, using the mode frequency of toothpaste use as reported by the parent. These analyses are considered secondary given toothpaste use is measured post-randomization and could potentially be influenced by the varnish the child received.

Additional regression analyses using the tooth surface as the unit of the analysis may be performed to evaluate the effect of tooth surface factors on the interventions. GEE methods will be used to account for the clustering of teeth and tooth surfaces within individual (Hardin & Hilbe, 2013). Analyses will be performed using R (The R Foundation for Statistical Computing, 2016; Version 3.3.0) and SAS (SAS Institute, Cary, NC, Version 9.4).

# 11.3.2 Analysis of Safety Data.

Adverse events (AEs) will be tabulated by treatment group, severity, and perceived relationship to investigational product. For each AE, treatment group comparisons regarding the occurrence of at least one event will be made using Fisher's exact tests. The comparisons will be repeated excluding all mild symptoms. Similar analyses will be performed after grouping AEs by body system using standard Medical Dictionary for Regulatory Activities (MedDRA) coding. Individual AEs will be listed, with particular attention paid to serious AEs.

# 11.3.3 Participant Disposition.

The frequency and reasons for withdrawal will be summarized by treatment group, as will the number of missed visits and missed treatment applications (compliance).

#### 12. Source Documents and Access to Source Data/Documents

The site will maintain appropriate medical and research records for this trial, in compliance with ICH E6, Section 4.9 and regulatory and institutional requirements for the protection of confidentiality of subjects.

#### **12.1 Primary Source Documents**

The Principal Investigator must maintain primary source documents supporting significant data for each subject in the subject's notes. During monitoring visits, the clinical site monitor will validate data in the CRF against these source data.

#### 12.2 CRF Worksheets

The site will be supplied with a set of forms-based schedule of activities and corresponding source document worksheets (SDW) that correspond to the case report form (CRF) for this study. The worksheets will serve as source documents for study observations. Additional source documentation for information not specifically included on the source document may be recorded on a separate document.

Access to the source documents should be limited to those working on the study. Access to the database will be restricted.

# 13. Ethics/Protection of Human Subjects

#### 13.1 Ethical Standard

This study will be conducted in accordance with the Good Clinical Practice (GCP) guidelines promulgated by the International Conference on Harmonization (ICH) and the Food and Drug Administration (FDA), and any applicable national and local regulations including FDA regulations under 21 CFR Parts 11, 50, 54, 56, 312 and 314.

The Principal Investigator will ensure that this study is conducted in full conformity with the principles set forth in The Belmont Report: Ethical Principles and Guidelines for the Protection of Human Subjects of Research, as drafted by the US National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research (April 18, 1979) and codified in 45 CFR Part 46 and/or the ICH E6; 62 Federal Regulations 25691 (1997).

#### 13.2 Institutional Review Board

The WCG IRB will review and approve the submission activities for the conduct of this protocol. The trial will not begin until the study has been approved by the WCG IRB, all required regulatory documentation is on file at both the site and the Principal Investigator and staff are trained on the protocol and data capture procedures.

#### 13.3 Amendments

The Principal Investigator will discuss any proposed protocol changes with the Sponsor and no modifications will be made without prior written approval and WCG IRB approval of the amended protocol, except where clinical judgment requires an immediate change for reasons of subject welfare. The WCG IRB will be informed of any amendments to the protocol or consent form, and approval (where and when appropriate) will be obtained before implementation.

#### **13.4 Informed Consent Process**

This study will be conducted in accordance with the provisions of 21 Code of Federal Regulations (CFR) Part 50.

In accordance with relevant regulations, a parent informed consent agreement explaining the procedures and requirements of the study, together with any potential hazards/risks must be read and/or explained to each parent/guardian. Each subject's parent or legal guardian will sign such an informed consent form. The subject's parent/guardian must be assured of the freedom to withdraw from participation in the study at any time.

It is the Principal Investigator's responsibility to make sure that the subject's parent/guardian understands what he or she is agreeing to and that written informed consent is obtained before the subject is involved in any protocol-defined procedures, including screening procedures. It is also the Principal Investigator's responsibility to retain the original signed consent forms and provide each subject's parent/guardian with a copy of the signed consent form.

As children will be enrolled in this study, the informed consent process will be documented in the form of permission from the parent or legal guardian in the parent permission form; child assent (affirmative agreement by a child to participate in research) will not be employed in this study.

# 13.5 Exclusion of Women, Minorities, and Children (Special Populations)

This study will enroll children aged 40 to 20 6 to 24 months. There will be no exclusion due to gender, race or ethnicity.

#### 13.6 Subject Confidentiality

The Principal Investigator must assure that the privacy of subjects, including their personal identity and personal medical information, will be maintained at all times. Personal medical information will always be treated as confidential. The parent/guardian's Authorization allows the Sponsor-Investigator to receive and review the subjects' protected health information that may be re-disclosed to any authorized representative of the Sponsor for review of subject medical records in the context of the study.

## 13.7 Study Discontinuation

At the completion of the study, study closeout procedures will be implemented.

# 14. Data Handling and Record Keeping

The Principal Investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

#### 14.1 Data Management Responsibilities

The Biostatistician will be responsible for all data collection procedures. The Data Management Plan includes, but is not limited to:

- Overview of data management processes utilized for study
- Universal data handling conventions
- Study-specific data handling conventions
- Coding dictionaries and practices
- Specifications for logic and edit checks
- External data handling practices
- Final study closeout activities
- Audit plans
- Sample CRF annotation
- Biostatistician contact information
- Section for tracking revisions to the plan
- Administrative report specifications

The Data Management Plan serves to document the practices and procedures deployed to promote consistent, efficient, and effective data management practices leading to the creation of a high-quality database ready for analysis. The plan serves as the authoritative source, documenting data management practices, and decisions that are agreed to with the Principal Investigator at the start of the study and as necessary updates are made during the conduct of the study.

Data will be transferred periodically from the study site to the University of Washington to prepare reports. At the close of the study, the locked database will be transferred to the Biostatistician for analysis.

The Biostatistician will be responsible for design of the randomization scheme, creation of analytical databases, and the statistical analysis plan.

#### **14.2 Data Capture Methods**

Clinical data (including AEs, concomitant medications, and expected adverse reactions data) will be entered into the study database by the Data Manager. This system is protected by 128-bit server certificates and utilizes authenticated, password-protected accounts for each site. The system is compliant with relevant FDA regulatory requirements per 21 CFR Part 11.

#### 14.3 Types of Data

Data for this study will include clinical assessments, safety, and outcome measures (e.g., expected adverse reactions). Safety data are contained in the clinical data set.

# 14.4 Timing/Reports

**Enrollments and study activity** (**protocol-specified reportable events**, as described in Section 9.6.1) reports will be generated as they occur to a pre-determined distribution list that includes the Principal Investigator and team.

**Clinical monitoring reports** will be generated periodically with electronic distribution to the PI and team. Per the Clinical Monitoring Plan, the clinical monitor reports include routine reports of aggregate, blinded adverse event data for ongoing review for potential trends, and adverse event and concomitant medication reports for the PI to review for standardization of coding.

**Safety monitoring reports** will be provided by the Biostatistician per the safety monitoring plan.

**Missing data, missing electronic signatures** of the Principal Investigator, and requests for **data clarification** reports will be generated to the site on a regular basis.

**Monitoring Visit Reports** will be generated after each clinical site monitoring visit, per the monitoring plan.

At the completion of the study, data will be securely transferred to the Biostatistician. Once the Biostatistician and the PI agree that all queries have been adequately resolved and the database has been deemed "clean", the database will be officially signed off and deemed locked. All permissions to make changes (append, delete, modify or update) the database are removed at this time.

All site personnel, Sponsor and staff will remain blinded as to treatment assignments until the conclusion of the entire study. A designated unblinded biostatistician will have access to the treatment assignments, and this individual will not communicate about study-related matters to any other staff involved in the study. The study code will be broken by the study-responsible statistician after all outstanding substantive data queries have been resolved.

#### 14.5 Study Records

### 14.5.1 Study File and Site Documents

The Principal Investigator should have the following study documents accessible to the Clinical Site Monitor during the study. These records are kept in the study office in Pohnpei.

- Signed Form FDA 1572
   This study will be conducted under the supervision and direction of the Principal Investigator listed in Section 1 of the Form FDA 1572. Sub-Investigators are listed in Section 6 of the Form FDA 1572. The study will be conducted at the address(es) listed in Section 3 of the Form FDA 1572.
- 2. Curriculum vitae for the Principal Investigator and all personnel listed on Form FDA 1572

The Principal Investigator is responsible for providing copies of the protocol and all other information relating to the preclinical and prior clinical experience, which were furnished to him/her, to all other study personnel who participate in this study. The Principal Investigator will discuss this information with them to assure that they are adequately informed regarding the investigational product and conduct of the study. The Principal Investigator must assure that all study staff members are qualified by education, experience and training to perform their specific responsibilities.

- 3. The signed IRB form/letter stating IRB approval of protocol, consent forms, and any other study materials (e.g., patient instruction materials, advertisement notices), documentation of the IRB composition, and all IRB correspondence including notification/approval of protocol amendments, notification of serious, unexpected, suspect adverse drug reactions to the IRB, and IRB notification of study termination
- 4. Training records
  Records of protocol-specific training will be maintained.
- 5. IRB-approved consent form
- 6. Signed protocol (and amendments, where applicable)
- 7. Signed parent/guardian permission forms
- 8. Copies of the completed source document worksheets
- 9. Delegation Log with names, signatures, initials, and functional role of all persons completing protocol assessments and providing back-up to the Principal Investigator.
- 10. Accountability of investigational product
- 11. Record of all monitoring visits by Clinical Site Monitor(s)
- 12. Copies of correspondence
- 13. Certificate for Human Subject Protection Program (HSPP) for each individual named on the Delegation Log who has direct subject contact
- 14. Copy of professional licensure/registration, as applicable, for each individual named on the Delegation Log, who has direct subject contact, ensuring licensure is in the locality in which the study will be conducted
- 15. The Principal Investigator must also retain adequate documentation, together with the subject's hospital/medical records, as the subject's source data for the study.

#### 14.5.2 Maintenance and Retention of Records

It is the responsibility of the Principal Investigator to maintain a comprehensive and centralized filing system of all relevant documentation. The Principal Investigator will be instructed to retain all study records required by federal regulations in a secure and safe facility with limited access for one of the following time periods based on notification from the Monitor.

The Principal Investigator will be instructed to consult with and provide advance written notice to the Monitor before disposal of any study records and to notify the Monitor of any change in the location, disposition, or custody of the study files. No

study document or image should be destroyed without prior written agreement between the Sponsor and the Principal Investigator.

Regulations require retention for:

- A period of at least two years after notification from the Sponsor that a U.S. NDA (New Drug Application) has been approved for the indication that was investigated or 15 years according to International Conference on Harmonization (ICH) guidelines.
- Or, if no NDA is filed or approved for such indication, a period of at least two
  years after the investigation is completed or discontinued, and the FDA (Food
  and Drug Administration) has been notified by the Sponsor.

#### 14.6 Protocol Deviations

A protocol deviation is accidental or unintentional changes to, or non-compliance with the research protocol that do not increase risk or decrease benefit or; do not have a significant effect on the subject's rights, safety or welfare; and/or on the integrity of the data. Deviations may result from the action of the subject, researcher, or research staff.

A deviation may be due to the research subject's non-adherence, or an unintentional change to or non-compliance with the research protocol on the part of a researcher. Examples of a deviation include: A rescheduled study visit; Failure to collect an ancillary self-report questionnaire; or Subject's refusal to complete scheduled research activities.

Protocol deviations will be recorded in the subject's file and log.

#### **14.7 Protocol Violations**

A protocol violation is any accidental or unintentional noncompliance with the WCG IRB approved protocol without prior approval requirements that may increase risk or decrease benefit, affects subjects' rights, safety, or welfare, or the integrity of the study data. The noncompliance may be either on the part of the subject, the Principal Investigator, or the study site staff. As a result of deviations, corrective actions are to be developed by the site and implemented promptly. These practices are consistent with ICH E6.

It is the responsibility of the site to use continuous vigilance to identify and report deviations within 5 working days of identification of the protocol deviation, or within 5 working days of the scheduled protocol-required activity. All deviations must be promptly reported to the Principal Investigator. The Study will maintain a database of violations that are not already documented in the clinical database. Corrective and preventive action plans will be documented to minimize recurrence of protocol violations, where applicable.

Protocol violations must be sent to the WCG IRB per WCG IRB guidelines. The Principal Investigator and staff are responsible for knowing and adhering to the WCG IRB requirements.

#### 15. Publication Policy

Following completion of the study, the Principal Investigator may submit for publication the results of this research in a scientific journal. The International Committee of Medical Journal Editors (ICMJE) member journals have adopted a trials-registration policy as a condition for publication. This policy requires that all clinical trials be registered in a public trials registry such as *ClinicalTrials.gov*, which is sponsored by the National Library of Medicine. Thus, the Sponsor will register this trial in the public trials registry, *ClinicalTrials.gov*.

#### 16. Literature References

American Academy of Pediatric Dentistry. Guideline on periodicity of examination, preventive dental services, anticipatory guidance/counseling, and oral treatment for infants, children, and adolescents. Pediatr Dent. 2013 Sep-Oct;35(5):E148-56.

American Academy of Pediatric Dentistry. Guideline on fluoride therapy. Pediatr Dent. 2013 Sep-Oct;35(5):E165-8.

Amin AS, Harrison RL, Benton TS, Roberts M, Weinstein P. Effect of povidone-iodine in children with extensive dental caries. Pediatr Dent 2004; 26: 5-10.

Berkowitz RJ, Koo H, McDermott M, Whelehan MT, Karp J, Billings RJ. Adjunctive chemotherapeutic suppression of mutans streptococci in the setting of severe early childhood caries. J Pub Health Dent 2009; 69(3):163-167.

Broadbent JM, Thomson WM, For debate: problems with the DMF index pertinent to dental caries data analysis. Community Dent Oral Epidemiol. 2005 December; 33(6):400–409.

Buchanan H, Niven N. Validation of a Facial Image Scale to assess child dental anxiety. Int J Paediatr Dent 2002; 12:47-52.

Caufield PW, Gibbons RJ. Suppression of Streptococcus mutans in the mouths of humans by a dental prophylaxis and topically-applied iodine. J Dent Res. 1979 Apr;58(4):1317-26.

Clark MB, Slayton RL, Section on Oral Health. Fluoride use in caries prevention in the primary care setting. Pediatrics 2014 Sept;134(3):626-633. doi:10.1542/peds.2014-1699

Furiga A1, Dols-Lafargue M, Heyraud A, Chambat G, Lonvaud-Funel A, Badet C. Effect of antiplaque compounds and mouthrinses on the activity of glucosyltransferases from

Streptococcus sobrinus and insoluble glucan production. Oral Microbiol Immunol. 2008 Oct;23(5):391-400.

Gao SS, Zhang S, Mei ML, Lo EC, Chu CH. Caries remineralization and arresting effect in children by professionally applied fluoride treatment – systematic review. BMC Oral Health. 2016 Feb 1;16(1):12.

Hardin JW, Hilbe JM. Generalized Estimating Equations, 2<sup>nd</sup> edition. Boca Raton FL: CRC Press. 2013.

Lin YS, Rothen ML, Milgrom P. Pharmacokinetics of lodine and Fluoride following Application of an Anticaries Varnish in Adults. JDR Clin Trans Res.2018 Jul;3(3):238-245.

Lopez L, Berkowitz RJ, Spiekerman C, Weinstein P. Topical antimicrobial therapy in the prevention of early childhood caries: a follow-up report. Pediatric Dent 24 2002: 204-206.

Milgrom P, Taves DM, Kim AS et al. Pharmacokinetics of fluoride in toddlers after application of 5% sodium fluoride dental varnish. Pediatrics 2014;134:e870–e874

Milgrom P, Tut OK, Mancl LA. Topical iodine and fluoride varnish effectiveness in the primary dentition: A guasi-experimental study. J Dent Child (Chic). 2011 Sep-Dec;78(3):143-7.

Milgrom P, Zero DT, Tanzer JM. An examination of the advances in science and technology of prevention of tooth decay in young children since the Surgeon General's Report on Oral Health. Acad Pediatr. 2009 Nov-Dec;9(6):404-9. doi: 10.1016/j.acap.2009.09.001.

Moyer VA, US Preventive Services Task Force. Prevention of dental caries in children from birth through age 5 years: US Preventive Services Task Force recommendation statement. Pediatrics. 2014 Jun;133(6):1102-11.

Schafer JL. Analysis of Incomplete Multivariate Data. London: Chapman & Hall, 1997.

Tam AI, Shemesh M, Wormser U, Sintov A, Steinberg D. Effect of different iodine formulations on the expression and activity of Streptococcus mutans glucosyltransferase and fructosyltransferase in biofilm and planktonic environments. J Antimicrob Chemother. 2006 May;57(5):865-71.

Tut OK, Milgrom P. Topical iodine and fluoride varnish combined is more effective than fluoride varnish alone for protecting erupting first permanent molars: a retrospective cohort study. J Public Health Dent 2010; (1): 1-4.

Weyant RJ, Tracy SL, Anselmo TT, Beltrán-Aguilar ED, Donly KJ, Frese WA, Hujoel PP, lafolla T, Kohn W, Kumar J, Levy SM, Tinanoff N, Wright JT, Zero D, Aravamudhan K, Frantsve-Hawley J, Meyer DM; American Dental Association Council on Scientific Affairs Expert Panel on Topical Fluoride Caries Preventive Agents. Topical fluoride for caries prevention: executive summary of the updated clinical recommendations and supporting systematic review. J Am Dent Assoc. 2013 Nov;144(11):1279-91.

# Phase 2 Efficacy & Safety Evaluation of Advantage Anti-Caries Varnish for Primary Prevention

Protocol # 2019-10-19


Zhan L, Featherstone JDB, Gansky SA, Hoover CI, Fujino T, Berkowitz RJ, DenBesten PK. Povidone iodine as an oral antiseptic in children with early childhood caries. J Pub Health Dent 2006 (3):174-179.

# 17. Addendum